CLINICAL TRIAL: NCT00461500
Title: Seretide 100 DK vs Flixotide 100 DK in IMT in Moderate Asthma in Adults on Static Lung Volumes (Mechanistic Study)
Brief Title: SERETIDE 100/50 bd (Twice Daily) Versus FLIXOTIDE 100 bd As Initial Maintenance Therapy In Moderate Asthma In Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAM108037
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Results first posted 2012-03-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Asthma
Keywords: persistent; moderate; asthma; adults; Initial; Maintenance; Therapy
MeSH Terms: conditions — Asthma; Lymphoma, Follicular | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

INTERVENTIONS:
Drug: Salmeterol xinafoate/fluticasone propionate combination — SFC 100
  Other Names: SERETIDE FLIXOTIDE
Drug: Fluticasone propionate — FP 100

SUMMARY:
This study will compare during 12 weeks, two treatment strategies for Initial Maintenance Therapy : fluticasone propionate alone or the salmeterol/fluticasone propionate combination in adults with moderate persistent asthma

DETAILED DESCRIPTION:
A multicentre randomised, double-blind, parallel-group study to compare the salmeterol/fluticasone propionate combination (SERETIDETM DISKUSTM 50/100) 50/100µg one inhalation twice daily with fluticasone propionate (FLIXOTIDETM DISKUSTM 100) 100µg one inhalation twice daily as initial maintenance therapy for 12 weeks in adults with persistent moderate asthma

ELIGIBILITY:
Inclusion criteria:

* male or female ≥ 18
* documented history of asthma
* reversibility FEV1 or PEF ≥ 12% (post 400µg salbu)
* moderate asthma (daily symptoms, daily rescue use, PEF = 60-80% predicted value)
* naive or ≥ 4weeks-free ICS (inhaled corticosteroids)

Exclusion criteria:

* respiratory disorder
* FEV1<60% predicted
* exacerbation/respiratory infection ≤ 4 weeks
* oral/parenteral/depot corticosteroids ≤ 6 months
* LABA/oral β2 agonist/ ALT/ theophylline ≤ 4 weeks
* smoker or former smoker ≥ 5 packs year

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- SFC (Salmeterol Xinafoate/Fluticasone Propionate Combination): Analysis population are all randomized subjects in this arm. 50/100ug - one inhalation twice daily
- FP (Fluticasone Propionate)100: Analysis population are all randomized subjects in this arm. 100ug - one inhalation twice daily
Period: Overall Study
Arm/Group | SFC (Salmeterol Xinafoate/Fluticasone Propionate Combination) | FP (Fluticasone Propionate)100
Started | 37 | 44
Completed | 30 | 38
Not Completed | 7 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Expired Drug Treatment | 1 | 1
Not completed — Study Stopped | 1 | 2
Not completed — Drug Treatment Misuse | 1 | 0
Not completed — No Longer Willing to Take Part in Study | 1 | 0
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined: Analysis population used in this arm is ITT (intent-to-treat) population (Randomised subjects who received at least one dose of study drug and with evaluation for at least one efficacy criteria).
- FP 100: Fluticasone Propionate.: Analysis population used in this arm is ITT population(Randomised subjects who received at least one dose of study drug and with evaluation for at least one efficacy criteria).
- Total: Total of all reporting groups
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate. | Total
Number analyzed (Participants) | 34 | 43 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (17.9) | 49.3 (19.3) | 48.4 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 13 | 18 | 31
Smoking Status [Number; unit: participants]
  Current Smoker | 5 | 4 | 9
  Ex-Smoker | 5 | 5 | 10
  Never Smoked | 24 | 34 | 58

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Morning Peak Expiratory Flow (PEF) Over Weeks 5-12
Description: Mini Wright Peak Flow Meter used to allow patients to monitor their asthma - Peak Flow (or PEF - peak expiratory flow) is a measurement of how fast you can blow out. When someone is well, their PEF is higher - when the airways are narrow (as in asthma), PEF is lower. Readings based on age, height and gender.
Time Frame: Baseline, Weeks 5-12
Population: Intent-to-Treat population are all randomized patients having received one study drug dose and had at least one complete efficacy assessment.
Measure: Mean (Standard Deviation); unit: Liters per minute (L/min)
Groups:
- SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined: 50/100ug - one inhalation twice daily
- FP 100: Fluticasone Propionate: 100ug - one inhalation twice daily
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 29 | 37
Liters per minute (L/min) | 59.21 (70.42) | 50.98 (71.05)
Statistical Analysis 1: Comparison: SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined vs FP 100: Fluticasone Propionate; Test type: Superiority or Other; p = 0.683, ANCOVA; Mean Difference (Net) = 7.23, 95% CI [-27.96 to 42.43], Standard Error of Mean 17.60 — mean difference = drug SFC 100 minus FP 100

2. Secondary Outcome: Change From Baseline in Pre-dose FEV1 (Forced Expiratory Volume in One Second) Through Week 12 (Using Last Observation Carried Forward [LOCF] Approach)
Description: FEV1 is the amount of air (in liters) you can blow out within one second. A spirometer is the device used to measure FEV1. With normal lungs and airways you can normally blow out most of the air from your lungs within one second. Age, height and gender is used to determine what is normal. Change from baseline could have been measured at any time during the study (up to Week 12), using the LOCF. In the LOCF approach, for each individual, missing values are replaced by the last observed value of that variable.
Time Frame: Baseline through Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Liters | 0.25 (0.37) | 0.11 (0.35)

3. Secondary Outcome: Change From Baseline in Pre-dose (Percent Predicted) FEV1 Through Week 12 (Using Last Observation Carried Forward [LOCF] Approach)
Description: Percent predicted is based on tables of normal values that use variables such as age, gender, and weight as a method of standardization. Spirometry results are expressed as a percentage, and are generally considered abnormal if less than 80 percent of the normal predicted value. Change from baseline could have been measured at any time during the study (up to Week 12), using the LOCF. In the LOCF approach, for each individual, missing values are replaced by the last observed value of that variable.
Time Frame: Baseline through Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Percentage predicted of FEV1
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Percentage predicted of FEV1 | 7.46 (12.34) | 4.97 (13.07)

4. Secondary Outcome: Change From Baseline in FEV1 Reversibility Through Week 12 (Using Last Observation Carried Forward [LOCF] Approach)
Description: Reversibility is calculated as the percentage improvement of FEV1 from baseline. Change from baseline could have been measured at any time during the study (up to Week 12), using the LOCF. In the LOCF approach, for each individual, missing values are replaced by the last observed value of that variable. Percent reversibility of FEV1 was calculated as follows: (Post-bronchodilator FEV1 - pre-bronchodilator FEV1)/pre-bronchodilator FEV1 x 100. A negative difference indicates less reversibility.
Time Frame: Baseline through Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 41
Percent change | -9.46 (16.47) | -4.05 (11.97)

5. Secondary Outcome: Change From Baseline in Pre-dose Forced Expiratory Vital Capacity (FVC) Through Week 12 (Using Last Observation Carried Forward [LOCF] Approach)
Description: FVC is the total amount of air that can forcibly be blown out after full inspiration, measured in liters. A spirometer is the device used to measure FVC. Age, height and gender is used to determine what is normal. Change from baseline could have been measured at any time during the study (up to Week 12), using the LOCF. In the LOCF approach, for each individual, missing values are replaced by the last observed value of that variable.
Time Frame: Baseline through Week 12
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Liters | 0.18 (0.44) | 0.14 (0.49)

6. Secondary Outcome: Change From Baseline (BL) in Pre-dose FEF 25-75% (Forced Expiratory Flow) Through Week 12 (Using Last Observation Carried Forward [LOCF] Approach)
Description: Forced Expiratory Flow 25-75% (measured by a spirometer) is the average flow (or speed) of air coming out of the lung during the middle portion of the expiration. Age, height, and gender is used to determine what is normal. Change from BL could have been measured at any time during the study (up to Week 12), using the LOCF (for each individual, missing values are replaced by the last observed value of that variable). Change from BL is measured as percentage of predicted value, with height, gender, age, and race as variables (percentage of predicted value at endpoint minus value at BL).
Time Frame: Baseline through Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Percentage of predicted value | 7.24 (24.07) | 4.28 (17.30)

7. Secondary Outcome: Number of Participants With at Least One Exacerbation During 12-Week Treatment Period
Description: Subjects will record exacerbations (defined as temporary PEF decrease, increase in salbutamol use) in a Daily Record Card (DRC). The number of events are categorized as those that showed a deterioration in asthma requiring administration of oral corticosteroids and/or a deterioration in asthma requiring emergency room visit and/or hospitalization (hosp.).
Time Frame: 12-Week Treatment Period (Week 1 through Week 12)
Population: Intent-to-Treat population.
Measure: Number; unit: Participants
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 34 | 43
Participants
  Any exacerbation (Exac.) | 1 | 5
  Exac. needing oral corticosteroids and/or hosp. | 0 | 0

8. Secondary Outcome: Number of Participants Who Achieved Well-Controlled Asthma During Weeks 5-12
Description: Well-controlled asthma is defined as 2 or more of the following: symptoms on no more than 2 days with symptom score of >1; no more than 2 days of rescue meds (maximum of 4 per week); >=80% predicted morning PEF. And no night time awakenings, exacerbations, emergency room visits, and treatment related adverse effects requiring a change to therapy. The number of participants who achieved "well-controlled" asthma at any time during Week 5-12 of the study period will be summarized by treatment groups. The difference between treatment groups will be assessed using logistic regression.
Time Frame: Weeks 5 -12
Population: Intent-to-Treat population.
Measure: Number; unit: Participants
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 29 | 35
Participants
  Yes | 13 | 11
  No | 16 | 24

9. Secondary Outcome: Median Number of Weeks to First Achieve Well-Controlled Asthma During Weeks 5-12
Description: Well-controlled asthma is defined as 2 or more of the following: symptoms on no more than 2 days with symptom score of >1; no more than 2 days of rescue meds (maximum of 4 per week); >=80% predicted morning PEF. And no night time awakenings, exacerbations, emergency room visits, and treatment related adverse effects requiring a change to therapy. The median number of weeks to first achieve "well-controlled" asthma during Week 5-12 of the study period will be summarized by treatment groups. The difference between treatment groups will be assessed using logistic regression.
Time Frame: Weeks 5 - 12
Population: Intent-to-Treat population.
Measure: Median (Full Range); unit: Weeks
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 34 | 43
Weeks | 3.1 [0.1 to 15.6] | 4.1 [0.1 to 14.1]

10. Secondary Outcome: Number of Participants Who Achieved Total-controlled Asthma During Weeks 5-12
Description: Totally-controlled asthma is defined as no daily symptoms, no night-time awakenings, no exacerbations, no rescue medication, no emergency visits, no treatment related adverse events resulting in change in asthma therapy, >=80% predicted PEF. The number of subjects who achieved "total-controlled" asthma at any time during Week 5-12 of the study period will be summarized by treatment groups. The difference between treatment groups will be assessed using logistic regression.
Time Frame: Weeks 5 - 12
Population: Intent-to-Treat population.
Measure: Number; unit: Participants
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 29 | 36
Participants
  Yes | 1 | 1
  No | 28 | 35

11. Secondary Outcome: Change From Baseline in Asthma Control Test (ACT) Score at Week 12
Description: 5 question test with various responses rating frequency of asthma events over 4-week period. Questions include occurrence of asthma affecting work/school; causing shortness of breath; symptoms (wheezing, coughing, shortness of breath, chest tightness, pain) wake you up at night; causing need for rescue medication; asthma control. Scale: 1=all of time, 2=most of time, 3=some of the time, 4=a little of the time, 5=none of the time. Possible ACT scores range from 5 to 25.
Time Frame: Baseline, Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Score on a scale | 5.64 (5.00) | 5.90 (4.81)

12. Secondary Outcome: ACT Score in Classes at Week 12
Description: Score is ranged from 5 (poor control) to 25 (complete control).
Time Frame: Week 12
Population: Intent-to-Treat population.
Measure: Number; unit: Particpants
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 42
Particpants
  < 15 score | 5 | 2
  15-19 score | 12 | 15
  >=20 score | 16 | 25

13. Secondary Outcome: Change From Baseline in Overall Asthma Quality of Life Questionnaire (AQLQ) Score at Week 12
Description: 7-point scale where 1=total impairment and 7=no impairment. Questions contain 32 items in four domains. Domains include Activity Limitation (11 items), Symptoms (12 items), Emotional Function (5 items), and Environmental Stimuli (4 items). 32 items produce one overall quality of life score. The 7 points scoring are different and depend on the item : they are the translation in French of the original questionnaire from Juniper. Possible AQLQ scores range from 1 to 7 (the mean of all the questions).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Number analyzed (Participants) | 33 | 41
Score on a scale | 0.99 (0.92) | 1.11 (1.02)

ADVERSE EVENTS:
Arm/Group | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/44
Other Adverse Events (participants affected / at risk) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | SFC 100: Salmeterol Xinafoate/Fluticasone Propionate Combined | FP 100: Fluticasone Propionate
Bronchitis (Infections and infestations) | 0/37 (0) | 2/44 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centres of a multi-centre trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.